CLINICAL TRIAL: NCT02546895
Title: Prospective Registration of Head and Neck Cancer Patients for Clinical Data and Tissue Collection
Brief Title: Prospective Registration of Head and Neck Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Han-Sin Jeong, Professor, Samsung Medical Center
Other Study IDs: 2015-06-132
Record Dates: First submitted 2015-08-11; First posted 2015-09-11 (Estimated); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer patients; clinical data; tissue collection; prospective registration; patients
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Serum
  2. Tissue specimen
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: chart review — The patient charts will be reviewed to determine pretreatment characteristics, treatment-related adverse events, time to progression and overall survival.
  Behavioral: Questionnaires Completion of 3 questionnaires 1 week before treatment(radiotherapy or chemotherapy) begins or been hospitalized for surgery the same day, 1 week after the end of treatment(expected average of 8 weeks), and again 3 months after treatment. It may take about 30 minutes to complete the questionnaires each time.
  Other Names: surveys

SUMMARY:
Head and neck cancers account for the sixth leading cause of cancers worldwide. The annual incidence of Head and neck cancers is more than 650,000 the patients each year. Head and neck cancers are associated with smoking, alcohol consumption, human papilloma virus (type 16 and 18) and previous exposure to radiation.

So far, most of clinical and research data about head and neck cancers, such as the etiology, pathogenesis, prognosis factors and associated factors, treatment outcomes, are from Western countries. However, due to various environmental factors, for example race, genetics, geographical factors, general hygiene and health care system differences, the possibility of differences of disease characteristics between Western and Asian people should be considered.

For several decades, there have been many studies about treatment modalities (surgery, chemotherapy, and radiation therapy), complications and side effects for head and neck cancers in the West. Many institutions tried to improve the survival rate and resolve the toxicity of chemotherapy and radiation treatment for head and neck cancer patients. However there has been little information about the characteristics of head and neck cancers, effectiveness of treatment (survival rate, recurrence, and complication rate), and prognosis, particularly in Korean as well as in Asian patients.

Therefore it is necessary to evaluate and analyze the features of head and neck cancers such as etiology, pathogenesis, risk factors, prognostic factors, treatment outcomes in a site specific cohort (South Korea) separately. It could be helpful to improve the treatment outcomes of head and neck cancers overall, to design race or site specific treatments for head and neck cancers, and to develop management strategy common in Asia as well as the West.

The purpose of this study is

1. To establish the prospective tumor registry about patient's information, treatment-related morbidities, treatment outcomes and quality of life, in addition to the prospective collection of patient samples (blood and tumor tissues).
2. To establish the predictive model for treatment outcomes and treatment-related morbidities.
3. To develop the biomarkers as predictive and/or prognostic factors.

DETAILED DESCRIPTION:
Review of medical records Medical records of enrolled patients will be reviewed to evaluate clinical characteristics, treatment-related adverse events, time to progression and overall survival.

Behavioral : Questionnaires 3 times : Prior to the 1 week before treatment(radiotherapy or chemotherapy) begins or been hospitalized for surgery the same day, 1 week after the end of treatment(expected average of 8 weeks), and again 3 months after treatment Other Names : Surveys

ELIGIBILITY:
Inclusion Criteria:

* Adults over 19 years-old
* Patients diagnosed as head and neck cancer histopathologically according to American Joint Committee on Cancer, Cancer staging manual, 7th edition at Samsung Medical Center:

  * Comprise a part of head and neck
  * Oral cavity
  * Pharynx
  * Larynx
  * Hypopharynx
  * Nasal cavity
  * Paranasal sinus
  * Nasopharynx
  * Salivary gland
  * Skin in the head and neck
* In case patients are diagnosed at other hospitals, it can be possible to register the tissue of cancer cell with Samsung medical center and confirm the diagnosis by pathologists of Samsung medical center.
* Histopathological type:

  * Squamous cell carcinoma
  * Malignant melanoma
  * Sarcoma and other carcinomas are included.
* Metastasis of Unknown Origin (MUO) at head and neck is included.
* Patients who receive a proper treatment as scheduled.
* Informed consents: patients who understand the purpose of study and are capable of giving a written consent.

Exclusion criteria:

* Patients who do not meet the requirements of inclusion criteria

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pathologically proven head and neck cancer patients, who are referred to Samsung Medical Center
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-09; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 years
  Revised RECIST guideline

SECONDARY OUTCOMES:
Identification of biomarkers of clinical significance (prognostic) | 5 years
  Biomarkers associated with treatment outcomes (HPV, Epidermal growth factor receptor, p53, p16, etc)
Number of participants with treatment-related morbidity | 5 years
  CTCAE protocol
Number of participants with treatment response | 5 years
  Number of participants with treatment response
Overall survival | 5 years
  Revised RECIST guideline
Scores of distress questionnaire | 1 week before treatment(radiotherapy or chemotherapy) begins or been hospitalized for surgery the same day, 1 week after the end of treatment(expected average of 8 weeks), and again 3 months after treatment
  QLQ HN43
Scores of support survey | 1 week before treatment(radiotherapy or chemotherapy) begins or been hospitalized for surgery the same day, 1 week after the end of treatment(expected average of 8 weeks), and again 3 months after treatment
  QLQ HN43
Quality of life score | 1 week before treatment(radiotherapy or chemotherapy) begins or been hospitalized for surgery the same day, 1 week after the end of treatment(expected average of 8 weeks), and again 3 months after treatment
  QLQ HN43

CONTACTS AND LOCATIONS:
Overall Officials: Han-Sin Jeong, M.D.Ph.D., Principal Investigator — Department of Otorhinolaryngology-Head and Neck Surgery, Sungkyunkwan University School of Medicine, Samsung Medical Center; Se-Hoon Lee, M.D.Ph.D., Principal Investigator — Department of Hemato-Oncology, Sungkyunkwan University School of Medicine, Samsung Medical Center; Dongryul Oh, M.D.Ph.D., Principal Investigator — Department of Radiation Oncology, Sungkyunkwan University School of Medicine, Samsung Medical Center; Chung-Hwan Baek, M.D.Ph.D., Study Chair — Department of Otorhinolaryngology-Head and Neck Surgery, Sungkyunkwan University School of Medicine, Samsung Medical Center; Young-Ik Son, M.D.Ph.D., Study Chair — Department of Otorhinolaryngology-Head and Neck Surgery, Sungkyunkwan University School of Medicine, Samsung Medical Center; Man Ki Chung, M.D.Ph.D., Study Chair — Department of Otorhinolaryngology-Head and Neck Surgery, Sungkyunkwan University School of Medicine, Samsung Medical Center; Young Chan Ahn, M.D.Ph.D., Study Chair — Department of Radiation Oncology, Sungkyunkwan University School of Medicine, Samsung Medical Center; Myung-Ju Ahn, M.D.Ph.D., Study Chair — Department of Hemato-Oncology, Sungkyunkwan University School of Medicine, Samsung Medical Center; Keunchil Park, M.D.Ph.D., Study Chair — Department of Hemato-Oncology, Sungkyunkwan University School of Medicine, Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Leemans CR, Braakhuis BJ, Brakenhoff RH. The molecular biology of head and neck cancer. Nat Rev Cancer. 2011 Jan;11(1):9-22. doi: 10.1038/nrc2982. Epub 2010 Dec 16. PMID 21160525
- [Background] Bonner JA, Harari PM, Giralt J, Azarnia N, Shin DM, Cohen RB, Jones CU, Sur R, Raben D, Jassem J, Ove R, Kies MS, Baselga J, Youssoufian H, Amellal N, Rowinsky EK, Ang KK. Radiotherapy plus cetuximab for squamous-cell carcinoma of the head and neck. N Engl J Med. 2006 Feb 9;354(6):567-78. doi: 10.1056/NEJMoa053422. PMID 16467544
- [Background] Posner MR, Hershock DM, Blajman CR, Mickiewicz E, Winquist E, Gorbounova V, Tjulandin S, Shin DM, Cullen K, Ervin TJ, Murphy BA, Raez LE, Cohen RB, Spaulding M, Tishler RB, Roth B, Viroglio Rdel C, Venkatesan V, Romanov I, Agarwala S, Harter KW, Dugan M, Cmelak A, Markoe AM, Read PW, Steinbrenner L, Colevas AD, Norris CM Jr, Haddad RI; TAX 324 Study Group. Cisplatin and fluorouracil alone or with docetaxel in head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1705-15. doi: 10.1056/NEJMoa070956. PMID 17960013
- [Background] Seiwert TY, Salama JK, Vokes EE. The chemoradiation paradigm in head and neck cancer. Nat Clin Pract Oncol. 2007 Mar;4(3):156-71. doi: 10.1038/ncponc0750. PMID 17327856
- [Background] Seiwert TY, Salama JK, Vokes EE. The concurrent chemoradiation paradigm--general principles. Nat Clin Pract Oncol. 2007 Feb;4(2):86-100. doi: 10.1038/ncponc0714. PMID 17259930
- [Background] Vermorken JB, Remenar E, van Herpen C, Gorlia T, Mesia R, Degardin M, Stewart JS, Jelic S, Betka J, Preiss JH, van den Weyngaert D, Awada A, Cupissol D, Kienzer HR, Rey A, Desaunois I, Bernier J, Lefebvre JL; EORTC 24971/TAX 323 Study Group. Cisplatin, fluorouracil, and docetaxel in unresectable head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1695-704. doi: 10.1056/NEJMoa071028. PMID 17960012
- [Background] Kumar B, Cordell KG, Lee JS, Worden FP, Prince ME, Tran HH, Wolf GT, Urba SG, Chepeha DB, Teknos TN, Eisbruch A, Tsien CI, Taylor JM, D'Silva NJ, Yang K, Kurnit DM, Bauer JA, Bradford CR, Carey TE. EGFR, p16, HPV Titer, Bcl-xL and p53, sex, and smoking as indicators of response to therapy and survival in oropharyngeal cancer. J Clin Oncol. 2008 Jul 1;26(19):3128-37. doi: 10.1200/JCO.2007.12.7662. Epub 2008 May 12. PMID 18474878
- [Background] Pignon JP, le Maitre A, Maillard E, Bourhis J; MACH-NC Collaborative Group. Meta-analysis of chemotherapy in head and neck cancer (MACH-NC): an update on 93 randomised trials and 17,346 patients. Radiother Oncol. 2009 Jul;92(1):4-14. doi: 10.1016/j.radonc.2009.04.014. Epub 2009 May 14. PMID 19446902
- [Background] Hitt R, Lopez-Pousa A, Martinez-Trufero J, Escrig V, Carles J, Rizo A, Isla D, Vega ME, Marti JL, Lobo F, Pastor P, Valenti V, Belon J, Sanchez MA, Chaib C, Pallares C, Anton A, Cervantes A, Paz-Ares L, Cortes-Funes H. Phase III study comparing cisplatin plus fluorouracil to paclitaxel, cisplatin, and fluorouracil induction chemotherapy followed by chemoradiotherapy in locally advanced head and neck cancer. J Clin Oncol. 2005 Dec 1;23(34):8636-45. doi: 10.1200/JCO.2004.00.1990. Epub 2005 Nov 7. PMID 16275937
- [Background] Bonner JA, Harari PM, Giralt J, Cohen RB, Jones CU, Sur RK, Raben D, Baselga J, Spencer SA, Zhu J, Youssoufian H, Rowinsky EK, Ang KK. Radiotherapy plus cetuximab for locoregionally advanced head and neck cancer: 5-year survival data from a phase 3 randomised trial, and relation between cetuximab-induced rash and survival. Lancet Oncol. 2010 Jan;11(1):21-8. doi: 10.1016/S1470-2045(09)70311-0. Epub 2009 Nov 10. PMID 19897418
- [Background] Hah, J. H. (2012). Personalized Treatment of Head and Neck Cancers and the Role of Head and Neck Surgeons. Korean Journal of Otorhinolaryngology-Head and Neck Surgery, 55(8), 471-475
- [Background] Glisson BS, Murphy BA, Frenette G, Khuri FR, Forastiere AA. Phase II Trial of docetaxel and cisplatin combination chemotherapy in patients with squamous cell carcinoma of the head and neck. J Clin Oncol. 2002 Mar 15;20(6):1593-9. doi: 10.1200/JCO.2002.20.6.1593. PMID 11896109
- [Derived] Kang D, Kim E, Choi N, Kim H, Cho J, Jeong HS. Pre-treatment quality of life in patients with salivary gland cancer in comparison with those of head and neck cancer patients. Qual Life Res. 2023 May;32(5):1493-1506. doi: 10.1007/s11136-022-03323-8. Epub 2022 Dec 13. PMID 36512301